CLINICAL TRIAL: NCT05846815
Title: Assessment of ARVO Web-based Software for Evaluating Attention-Deficit/Hyperactive Disorder (ADHD) Symptoms in Children. Prospective, Controlled Clinical Investigation
Brief Title: Assessment of ARVO Web-based Software for Evaluating Attention-Deficit/Hyperactive Disorder (ADHD) Symptoms in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peili Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Arvo-001
Record Dates: First submitted 2023-04-19; First posted 2023-05-06 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, case control clinical investigation. Comparison of groups.
  Equivalence study. Intervention model: cross-over assignment both groups are given both ARVO and Conners Continuous Performance Test 3rd Edition™ (CPT 3) tests.
  Allocation: Propensity matching is used to ensure inter-group homogeneity in background variable with possible interaction effect to ARVO and CPT 3 score. Propensity matching: age and sex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TD (Experimental): Children of 8-13 years of age without any neuropsychiatric diagnose (typically developed)
  Interventions: Device: ARVO 2.0 WEB; Other: Conners Continuous Performance Test 3rd Edition™ (CPT 3)
- ADHD (Experimental): Children of 8-13 years of age with previously diagnosed ADHD symptoms
  Interventions: Device: ARVO 2.0 WEB; Other: Conners Continuous Performance Test 3rd Edition™ (CPT 3)

INTERVENTIONS:
Device: ARVO 2.0 WEB — Medical device software where the subject navigates in a virtual apartment, with the goal of performing the tasks given by a cartoon dragon character. The child is asked to perform the subtasks in the given order, except for the subtasks to be completed at a certain time or after a certain sound cue, but the completion order does not influence the scoring. One task scenario lasts until all subtasks are correctly performed or until the time limit of 60 s is reached.
  The classification whether the subject belong to typically developed population is based on quantitative neurological performance indicators produced during the game. However, even if the activity performed is differential diagnostics, ARVO does not create any medical diagnosis. It shall be also noted that in the present clinical investigation, the interpretation of the results regarding child's ADHD susceptibility is not performed.
Other: Conners Continuous Performance Test 3rd Edition™ (CPT 3) — Subjects are required to respond by pressing the spacebar or the appropriate key on the mouse when any letter other than the letter "X" appears on the monitor. The Conners CPT 3 presents 14-minute, 360 scored stimuli trials (i.e., individual letters) on the screen, with 1, 2, or 4 sec. between the presentation of letters (i.e., the interstimulus interval; ISI). The 360 trials are divided into 6 blocks, with 3 sub-blocks each consisting of 20 trials. Each block lasts approximately 2 min and 20 sec. Scores and Score Dimensions of Attention Measured: Inattentiveness, Impulsivity, Sustained Attention and Vigilance. The Conners CPT 3 produces computer-generated reports that describe the respondent's performance.
  It shall be also noted that in the present clinical investigation, the interpretation of the results regarding child's ADHD susceptibility is not performed

SUMMARY:
Clinical investigation is aimed to assess the performance and safety of web-based ARVO 2.0, for evaluating possible Attention-Deficit/Hyperactive Disorder (ADHD) symptoms in children. Possible ADHD symptoms are recorded by using specific predetermined neurocognitive performance indicators (NPI's), derived during/from the game.

Results of ARVO are compared to the Conners Continuous Performance Test 3rd Edition™ (CPT 3) that is a task-oriented, automated 14-minute computerized assessment of attention-deficit (AD) related problems in individuals aged 8 years and older.

Performance and safety of ARVO and CPT 3 are compared in two clinical investigation populations, 8-13 years old ADHD children and typically developing (TD) children of the same age. Test are performed by the subject while monitoring adult supervises safety of the use.

ELIGIBILITY:
Inclusion Criteria:

ADHD group

The Inclusion criteria:

1. Signed informed consent (by guardian and a child)
2. Age of 8-13 at the time of consent
3. ADHD set by a licensed physician
4. Native language Finnish / Fluent Finnish language

TD group

The Inclusion criteria:

1. Signed informed consent (by guardian and child)
2. Age of 8-13 at the time of the consent
3. Native language Finnish / Fluent Finnish language

Exclusion Criteria:

ADHD group

1. Any diseases of the nervous system (ICD-10, G00-G99)
2. Mental and behavioural disorders due to psychoactive substance use (F10-F19)
3. Schizophrenia, schizotypal and delusional disorders (F20 - F29)
4. Acute severe depression or mania / hypomania (F30, F32, F33)
5. Phobic anxiety disorders, other anxiety disorders, obsessive-compulsive disorder (F40-F42)
6. Severe mental retardation (F72)
7. Disorders of psychological development (F80, F81, F83, F84)
8. Medication taken for ADHD (methylphenidate, lisdexamfetamine) on the test day (24 hour wash out)
9. Atomoxetine, guanfacine
10. Hearing or vision diagnosis (H90 Bilateral hearing loss, H53 Visual disturbances, H54 Blindness and low vision) Diagnosis search completeness criteria: Diagnosis present/absent in patient registry Kanta.

TD group

1. Set ADHD diagnosis.
2. Ongoing process related to setting an ADHD diagnosis, according to guardian's questionnaire.
3. Any diseases of the nervous system (ICD-10, G00-G99)
4. Mental and behavioural disorders due to psychoactive substance use (F10-F19)
5. Schizophrenia, schizotypal and delusional disorders (F20 - F29)
6. Acute severe depression or mania / hypomania (F30, F32, F33)
7. Phobic anxiety disorders, other anxiety disorders, obsessive-compulsive disorder (F40-F42)
8. Severe mental retardation (F72)
9. Disorders of psychological development (F80, F81, F83, F84)
10. Hearing or vision diagnosis (H90 Bilateral hearing loss, H53 Visual disturbances, H54 Blindness and low vision)

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
ARVO and CPT 3 neuropsychiatric indicators (NPIs) | At Visit 1 test event (four weeks after V0 enrollment)
  To confirm that ARVO is equivalent to (CPT 3) regarding predictive validity (AUC)
Children SSQ score | At Visit 1 (four weeks after V0 enrollment) immediately upon completed ARVO test
  To confirm that ARVO is safe as defined by Simulator Sickness Score (SSQ) value 0, 1, or 2.

SECONDARY OUTCOMES:
ARVO and CPT 3 neuropsychiatric indicators (NPIs) | Visit 1 test event (four weeks after V0 enrollment)
  To confirm that ARVO is equivalent to CPT 3 regarding individual NPIs ability to differentiate ADHD and TD groups
ARVO NPIs mean score and ADHR-RS for parent score | Visit 1 test event (four weeks after V0 enrollment)
  To confirm that ARVO is equivalent to ADHD-RS regarding concurrent validity (correlation)
Smileyometer and Fun Sorter | Visit 1 test event (four weeks after V0 enrollment)
  To confirm that ARVO is superior to CPT 3 regarding use experience

CONTACTS AND LOCATIONS:
Overall Officials: Sami Leppämäki, MD, PhD, Principal Investigator — Pro Neuron Oy
Locations (1):
- Pro Neuron Oy, Espoo, Finland

IPD SHARING:
Plan to Share IPD: Yes
By utilizing the data collected in this clinical investigation, the suitability of the web browser version of ARVO test to identify ADHD will be evaluated by metrics including number of correctly performed tasks, task efficiency, navigation efficiency, number of functions, and mouse movement speed. Additionally, it will be evaluated whether other metrics that are central to the assessment of ADHD can be identified from the collected data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2024-2030
Access Criteria: Scientific research as defined in the Clinical Investigation Plan and supporting documents.